CLINICAL TRIAL: NCT03037762
Title: Findings and Side-effects of Flexible Endoscopic Evaluation of Swallowing - the FEES-Registry
Acronym: FEES-Registry
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: 01072014
Record Dates: First submitted 2017-01-12; First posted 2017-01-31 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Neurogenic Dysphagia; Flexible Endoscopic Evaluation of Swallowing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Flexible Endoscopic Evaluation of Swallowing

SUMMARY:
Neurogenic dysphagia is one of the most frequent and prognostically relevant neurological deficits in a variety of disorders, such as stroke, parkinsonism and advanced neuromuscular diseases. Flexible endoscopic evaluation of swallowing (FEES) is now probably the most frequently used tool for objective dysphagia assessment in Germany. It allows evaluation of the efficacy and safety of swallowing, determination of appropriate feeding strategies and assessment of the efficacy of different swallowing manoeuvres. The literature furthermore indicates that FEES is a safe and well-tolerated procedure. The FEES-Registry aims at evaluating findings and side effects of FEES in a heterogeneous collective of patients with neurogenic dysphagia.

ELIGIBILITY:
Inclusion criteria:

* suspected neurogenic dysphagia
* Patients being scheduled for a FEES
* written informed consent

Exclusion criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected neurogenic dysphagia
Sampling Method: Non-Probability Sample
Enrollment: 2401 (Actual)
Dates: Start 2014-10; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
FEES-related side effects - 1. systolic blood pressure increase | during the procedure
  Systolic blood pressure will be measured directly prior, during and after the procedure. The initial value will be compared to the highest blood pressure value measured during/directly after the procedure.
FEES-related side effects - 2. Oxygen saturation decline | during the procedure
  Oxygen saturation will be measured directly prior, during and directly after the procedure. The initial value will be compared to the lowest value measured during/directly after the procedure.
FEES-related side effects - 3. Heart rate decrease | during the procedure
  Heart rate will be measured directly prior, during and directly after the procedure. The initial value will be compared to the lowest value measured during/directly after the procedure.
FEES-related side effects - 4. Nose bleed | during the procedure
  Number of patients with nose bleed during the procedure
FEES-related side effects - 5. Laryngospasm | during the procedure
  Number of patients with laryngospasm during the procedure
FEES-related side effects - 6. Decreased level of consciousness | during the procedure
  Number of patients with a decline in consciousness during the procedure (measured with the Richmond agitation and sedation scale)
Patients subjective FEES-related discomfort | during the procedure
  Number of patients with procedure related discomfort measured with a 4 point scale ranging from 1=no discomfort to 4=extremely painful sensation during the procedure

SECONDARY OUTCOMES:
Changes of dietary status after FEES | immediately prior and immediately after the procedure
  Dietary status will be assessed directly prior to the procedure and immediately thereafter. Dietary status will be assessed with the Functional Oral Intake Scale (FOIS scale).

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Dziewas, MD, Principal Investigator — University Hospital Muenster, Department of Neurology, Germany
Locations (1):
- University Hospital, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dziewas R, Auf dem Brinke M, Birkmann U, Brauer G, Busch K, Cerra F, Damm-Lunau R, Dunkel J, Fellgiebel A, Garms E, Glahn J, Hagen S, Held S, Helfer C, Hiller M, Horn-Schenk C, Kley C, Lange N, Lapa S, Ledl C, Lindner-Pfleghar B, Mertl-Rotzer M, Muller M, Neugebauer H, Ozsucu D, Ohms M, Perniss M, Pfeilschifter W, Plass T, Roth C, Roukens R, Schmidt-Wilcke T, Schumann B, Schwarze J, Schweikert K, Stege H, Theuerkauf D, Thomas RS, Vahle U, Voigt N, Weber H, Werner CJ, Wirth R, Wittich I, Woldag H, Warnecke T. Safety and clinical impact of FEES - results of the FEES-registry. Neurol Res Pract. 2019 Apr 26;1:16. doi: 10.1186/s42466-019-0021-5. eCollection 2019. PMID 33324882